CLINICAL TRIAL: NCT04122196
Title: Perioperative Pregabalin as Part of a Multimodal Treatment Plan for Ureteral Stent Symptoms After Ureteroscopy: a Randomized Controlled Trial
Brief Title: Perioperative Pregabalin in Ureteroscopy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Eliza DeFroda, Assistant Professor, Urology, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017676
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Kidney Stone; Pain, Postoperative; Addiction; Opioid Use
MeSH Terms: conditions — Kidney Calculi; Pain, Postoperative; Behavior, Addictive | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pregabalin 300mg (Experimental): Patient will receive a compounded version of 300mg pregabalin PO approximately one hour before surgery.
  Interventions: Drug: Pregabalin 300mg
- Placebo (Placebo Comparator): Patient will receive a compounded version of inactive placebo PO approximately one hour before surgery.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Pregabalin 300mg — Patient will receive a compounded version of 300mg pregabalin PO approximately one hour before surgery.
  Other Names: Lyrica
  Arms: Pregabalin 300mg
Drug: Placebo oral tablet — Patient will receive a compounded version of inactive placebo PO approximately one hour before surgery.
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blinded study examining the use of perioperative pregabalin in ureteroscopy with stent placement. Ureteroscopy is typically performed for kidney or ureteral stones, but may be performed for other reasons such as for the diagnosis and possible treatment of certain kinds of cancers. As part of the same surgery, a ureteral stent is often placed. The surgery and the stent can cause discomfort, and patients may receive narcotic pain medicine. In other surgeries, a single dose of pregabalin, around one hour before surgery has been shown to decrease the need for pain medication after the surgery. This work will test whether this is true in ureteroscopy by giving eligible patients who agree to participate either pregabalin or a placebo shortly before surgery then examining how much pain medication they use after surgery. A placebo is an inactive medication. Neither the study participant nor the study staff will know who received pregabalin and who received placebo until after the study is over. For completing surveys, patients will receive compensation for their time in the form of gift certificates.

DETAILED DESCRIPTION:
The prevalence of urolithiasis is greater than 8% and increasing in the United States. For those who require surgery, ureteroscopic treatment is common, representing >120,000 procedures yearly in the United States. This does not include ureteroscopy for other, including diagnosis of structural anomaly and diagnosis and management of ureteral and renal pelvic tumors. Frequently, a ureteral stent is placed intraoperatively. There is post-operative pain in around 80% of patients, and 12% of those undergoing ureteroscopy will have an emergency department visit in the first 30 post-operative days, typically for stent related symptoms or post procedural pain. Aside from the short-term repercussions of ureteroscopy with stent placement there are long-term issues related to pain and the treatment thereof. Recent evidence suggests that approximately 6% of opioid naïve patients who undergo ureteroscopy will become new persistent opioid users.

A single perioperative dose of pregabalin has been shown in many surgical contexts to have analgesic, anxiolytic, and opioid sparing effects. A common regimen employed in the literature is a single preoperative dose of 300mg PO pregabalin 1hr before induction of anesthesia. Pregabalin is a well-tolerated gabapentinoid medication with temporary cognition/coordination changes being the most common side effects. There is currently no standard of care for the use of perioperative gabapentinoid medication in ureteroscopy. A pilot was performed looking at such use that demonstrated the safety of this use and the feasibility of studying this at our institution.

In this work, the efficacy and safety of perioperative pregabalin in ureteroscopy with stent placement will be evaluated by executing a prospective, double blind, randomized, placebo-controlled trial for the use of perioperative pregabalin in the management of post-ureteroscopy symptoms, with the hypothesis that this treatment is safe and efficacious. Emphasis will be placed on patient-centered outcomes, especially those related to opioid sparing effects, mainly within the first 30 days after the surgery and extending out to one year.

The study will be powered with an 80% probability to detect a 10% difference in the primary outcomes. It will also assume a loss to follow up rate of 50%. This will require approximately 200 total subjects with a planned 1:1 placebo to active treatment enrollment ratio. The necessary enrollment can be accomplished in 11 months, allowing for 30 days of follow up within the funding period.

The final goal of this project will be at least one paper in a top urology journal. This will contribute to the literature by helping to inform urologists and anesthesiologists on the efficacy and safety of perioperative pregabalin for ureteroscopy with stent placement and will provide data regarding opioid sparing management after ureteroscopy. Opioid related issues abound nationwide and are evident in Missouri. This study has the potential to influence opioid use both in this state and nationwide as it relates to this frequently performed procedure.

ELIGIBILITY:
Subject Inclusion:

* Age >= 18 years
* Subject Population Undergoing elective ureteroscopy with stent placement at University of Missouri Hospital and affiliated facilities

Subject Exclusion:

* Renal insufficiency (eGFR < 60 mL/minute/1.73 m2)
* Chronic indwelling ureteral stent (>30 days in the previous year)
* Chronic opioid use
* History of opioid abuse
* Chronic gabapentinoid use
* History of gabapentinoid abuse
* Plan for inpatient hospitalization
* Pregnancy
* Inability of the patient to consent for themselves in English
* Allergy to gabapentinoid
* Liver failure or hepatic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katie Murray, DO, Principal Investigator — Assistant Professor
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

REFERENCES:
- [Background] Ahles TA, Ruckdeschel JC, Blanchard EB. Cancer-related pain--II. Assessment with visual analogue scales. J Psychosom Res. 1984;28(2):121-4. doi: 10.1016/0022-3999(84)90004-7. PMID 6737324
- [Background] Watson YI, Arfken CL, Birge SJ. Clock completion: an objective screening test for dementia. J Am Geriatr Soc. 1993 Nov;41(11):1235-40. doi: 10.1111/j.1532-5415.1993.tb07308.x. PMID 8227899

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pregabalin 300mg | Placebo
Started | 59 | 59
Completed | 59 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin 300mg | Placebo | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [32 to 59] | 57 [41 to 69] | 49 [36 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 31 | 67
  Male | 23 | 28 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 59 | 59 | 118
Total oral morphine equivalents in 30 days prior [Median (Inter-Quartile Range); unit: mg] | 8 [0 to 143] | 0 [0 to 100] | 4 [0 to 130]
Preoperative alpha blocker [Count of Participants; unit: Participants] | 27 | 28 | 55
First ureteroscopy [Count of Participants; unit: Participants] | 48 | 46 | 94
Prestented [Count of Participants; unit: Participants] | 23 | 15 | 38
Preoperative Watson Clock Test Score [Median (Inter-Quartile Range); unit: units on a scale] — This score is based on the scoring method described in Watson et al 1993. Higher scores demonstrate more errors. A clock is drawn. This is divided into quadrants. For errors in quadrants 1-3 (clock 12-8), a score of 1 is assigned. For errors in quadrant 4, a score of 4 is assigned. The scores are summed. Total scores range from 0 to 7 with 7 representing significant impairment (worst) and 0 representing no impairment (best).
  units on a scale | 2 [0 to 2] | 2 [0 to 2] | 2 [0 to 2]
Preoperative visual analogue scale of pain [Median (Inter-Quartile Range); unit: units on a scale] — This was a visual analogue scale of pain as described in Ahles et al 1984. The patients were given a paper with a 10cm horizontal line on it. On the left was marked "No pain" and on the right "Worst pain imaginable". The patients were then asked to mark a vertical line along the 10cm line that indicated where their pain was. The score is the number of centimeters from the left. 0 is minimum (best). 10 maximum (worst).
  units on a scale | 0.6 [0 to 3.5] | 0.5 [0 to 2.2] | 0.6 [0 to 2.7]
Stone location [Count of Participants; unit: Participants]
  Renal | 18 | 13 | 31
  Ureteral | 38 | 39 | 77
  None | 3 | 7 | 10
Laterality [Count of Participants; unit: Participants] — Population: Information not available for one participant
  Participants
    number analyzed (Participants) | 59 | 58 | 117
    Bilateral | 5 | 6 | 11
    Left | 32 | 30 | 62
    Right | 22 | 22 | 44
Stented at ureteroscopy [Count of Participants; unit: Participants] — While technically after randomization/medication administration, this characteristic is unlikely to depend on the randomization/medication administration and instead should be considered a baseline characteristic when evaluating the primary endpoint (post operative pain).
  Participants | 45 | 48 | 93
Sheath [Count of Participants; unit: Participants] — Sheath used during ureteroscopy.
  While technically after randomization/medication administration, this characteristic is unlikely to depend on the randomization/medication administration and instead should be considered a baseline characteristic when evaluating the primary endpoint (post operative pain).
  Participants | 35 | 31 | 66
Procedure length [Median (Inter-Quartile Range); unit: minutes] — While technically after randomization/medication administration, this characteristic is unlikely to depend on the randomization/medication administration and instead should be considered a baseline characteristic when evaluating the primary endpoint (post operative pain).
  minutes | 37 [21 to 57] | 38 [25 to 57] | 38 [22 to 57]
In-facility belladonna-opium suppository [Count of Participants; unit: Participants] — While technically after randomization/medication administration, this characteristic is unlikely to depend on the randomization/medication administration and instead should be considered a baseline characteristic when evaluating the primary endpoint (post operative pain).
  Participants | 14 | 11 | 25
In-facility non-steroidal anti-inflammatory drug [Count of Participants; unit: Participants] — While technically after randomization/medication administration, this characteristic is unlikely to depend on the randomization/medication administration and instead should be considered a baseline characteristic when evaluating the primary endpoint (post operative pain).
  Participants | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale of Pain Score
Description: This was a visual analogue scale of pain as described in Ahles et al 1984. The patients were given a paper with a 10cm horizontal line on it. On the left was marked "No pain" and on the right "Worst pain imaginable". The patients were then asked to mark a vertical line along the 10cm line that indicated where their pain was. The score is the number of centimeters from the left. 0 is minimum (best). 10 maximum (worst).
Time Frame: 1 hour after arrival to post anesthesia care unit
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Pregabalin 300mg | Placebo
Number analyzed (Participants) | 59 | 59
units on a scale | 3.7 [1.5 to 6.3] | 2.0 [0.6 to 4.2]

2. Secondary Outcome: Oral Morphine Equivalents of Opioids Prescribed
Time Frame: Within the first 30 days post-operation
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Pregabalin 300mg | Placebo
Number analyzed (Participants) | 59 | 59
mg | 60 [13 to 90] | 50 [0 to 60]

3. Secondary Outcome: Proportion of Patients With Narcotic Prescription
Time Frame: Within the first 30 days post-operation
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin 300mg | Placebo
Number analyzed (Participants) | 59 | 59
Participants | 44 | 35

4. Secondary Outcome: Number of Unplanned Healthcare Interactions
Description: Unplanned healthcare interactions include unplanned visits, emergency room visits, admissions to the hospital, and phone calls
Time Frame: Within the first 30 days post-operation
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin 300mg | Placebo
Number analyzed (Participants) | 59 | 59
Participants | 8 | 16

5. Secondary Outcome: Number of Serious Adverse Events
Description: Composite of unplanned serious adverse events including intensive care unit stay and death
Time Frame: Within the first 30 days post-operation
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin 300mg | Placebo
Number analyzed (Participants) | 59 | 59
Participants | 0 | 0

6. Secondary Outcome: Watson Clock Drawing Test Score
Description: This score is based on the scoring method described in Watson et al 1993. Higher scores demonstrate more errors. A clock is drawn. This is divided into quadrants. For errors in quadrants 1-3 (clock 12-8), a score of 1 is assigned. For errors in quadrant 4, a score of 4 is assigned. The scores are summed. Total scores range from 0 to 7 with 7 representing significant impairment (worst) and 0 representing no impairment (best).
Time Frame: 1 hour after arrival to post anesthesia care unit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin 300mg | Placebo
Number analyzed (Participants) | 59 | 59
units on a scale | 1.8 (2.1) | 1.8 (2.2)

7. Other Pre Specified Outcome: In-facility Oral Morphine Equivalents
Time Frame: Day of surgery
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Pregabalin 300mg | Placebo
Number analyzed (Participants) | 59 | 59
mg | 38 [30 to 63] | 35 [30 to 48]

8. Other Pre Specified Outcome: Nausea/Vomiting in PACU
Time Frame: In post anesthesia care unit (usually approximately 1 hour post op)
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin 300mg | Placebo
Number analyzed (Participants) | 59 | 59
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 30 days after procedure
Description: We prospectively collected this using a questionnaire. We also performed chart reivew.
Arm/Group | Pregabalin 300mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT04122196/Prot_001.pdf
  • Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT04122196/SAP_000.pdf